CLINICAL TRIAL: NCT01481883
Title: A Randomised Controlled Trial of Selective Estrogen Receptor Modulators (SERMs) - A Potential Treatment for Psychotic Symptoms of Schizophrenia in Men?
Brief Title: Selective Estrogen Receptor Modulators (SERMs) - A Potential Treatment for Psychotic Symptoms of Schizophrenia in Men?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Selective Estrogen Receptor Modulators (SERMs) - A Potential Treatment for Psychotic Symptoms of Schizophrenia in Men?, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 486/11
Record Dates: First submitted 2011-11-16; First posted 2011-11-30 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Mental Illness; SERM; Raloxifene
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Raloxifene Hydrochloride; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raloxifene Hydrochloride 120mg oral per day (Experimental): 120mg raloxifene plus antipsychotic drug
  Interventions: Drug: Raloxifene Hydrochloride
- Placebo tablet - one per day (Placebo Comparator): Lactose pill plus antipsychotic medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raloxifene Hydrochloride — 120mg daily - 1 capsule daily for 12 week trial
  Other Names: Evista; Raloxifene
  Arms: Raloxifene Hydrochloride 120mg oral per day
Drug: Placebo — 1 capsule daily for 12 week trial
  Other Names: Lactose
  Arms: Placebo tablet - one per day

SUMMARY:
The aim of this project is to investigate the effect of Raloxifene 120mg in men with schizophrenia. This trial will adopt a 12 week randomised controlled model.

Hypotheses 1: That the men receiving adjunctive selective estrogen receptor modulators (SERM) will have a significantly greater reduction in psychosis symptoms over the course of the study than men receiving adjunctive placebo.

Hypotheses 2: That the men receiving adjunctive SERM will have a significantly greater improvement in cognitive function than men receiving adjunctive placebo

DETAILED DESCRIPTION:
With the recent advent of selective estrogen receptor modulators (SERMS), such as raloxifene hydrochloride, there is the potential to harness the positive estrogenic effect on central nervous system (CNS) neurotransmitter systems. While the CNS effects of raloxifene have not been fully studied, its actions are mediated through binding to estrogen receptors and can thereby regulate gene expression that is ligand, tissue or gene specific. By inference then, raloxifene would be expected to impact on dopamine and serotonin pathways in a similar fashion to unconjugated estrogen.

This study aims to examine the impact of adjunctive SERM (120mg oral Raloxifene daily) treatment on the psychopathology and cognition of men with schizophrenia and related disorders

ELIGIBILITY:
Inclusion Criteria:

* Physically well
* DSM-IV diagnosis of schizophrenia, schizoaffective or schizophreniform
* 18- 45 years
* Able to give informed consent
* PANSS total score > 60 (1 - 7 scale) and a score of 4 (moderate) or more on two or more of the following PANSS items: delusions, hallucinatory behaviour, conceptual disorganization or suspiciousness

Exclusion Criteria:

* Patients with known abnormalities in the hypothalamo-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, active or past history of a venous thromboembolic event.
* Patients with any significant unstable medical illness such as epilepsy and diabetes or known active cardiac, renal or liver disease; presence of illness causing immobilization.
* Patients whose psychotic illness is directly related to illicit substance use or who have a history of substance abuse or dependence during the last six months, or consumption of more than 30gm of alcohol (three standard drinks) per day
* Smoking more than 20 cigarettes per day.
* Use of any form of estrogen, progestin or androgen as hormonal therapy, or antiandrogen including tibolone or use of phytoestrogen supplements as powder or tablet.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 12 week follow up in PANSS-positive and negative syndrome scale | baseline, week2, week4, week 6, week 8, week 10, week 12
  Positive and Negative Symptom Schedule (PANSS): The PANSS will be performed at baseline and at weeks 2,4,6,8,10 and 12. The PANSS consists of a Positive Scale (7 positive symptom constructs), a Negative Scale (7 negative symptom constructs) and a General Psychopathology Scale (16 symptom constructs). For each patient, the scale will be administered by the same trained rater. The PANSS provides a well standardised method of evaluating and monitoring psychotic symptoms. The rater is trained and recertified against an internationally recognised "gold standard".

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS): | baseline, week2, week4, week 6, week 8, week 10, week 12
  Montgomery Asberg Depression Rating Scale (MADRS): The MADRS will be performed at baseline, then at weeks 2,4,6,8,10 and 12. Many patients with schizophrenia have co-existing depression, hence monitoring of depression is important.
MATRICS Consensus Cognitive Battery | Baseline, week 12
  MATRICS Consensus Cognitive Battery (MCCB): The MATRICS test battery will be conducted at baseline and at study completion to quantify changes in cognitive functioning. This standardized battery assess the key separable cognitive deficits in schizophrenia and has a high test-retest reliability. The MATRICS comprises 7 Domains of which we will be assessing speed of processing, working memory, verbal learning, visual learning and reasoning and problem solving.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, week 12
  A neuropsychological test battery will be conducted at baseline and study completion to quantify changes in cognitive functioning. The RBANS comprises 12 subtests that are used to calculate five index scores (Immediate Memory; Visuospatial/Constructional; Language; Attention and Delayed Memory) and a total score. There are alternate forms to be used at each time point to avoid practice effects. The inclusion of the RBANS will allow direct comparisons in cognitive functioning with our other estrogen trials.

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, Phd,FRANZCP, Principal Investigator — Monash Alfred Psychiatry Research Centre
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Kulkarni J, de Castella A, Headey B, Marston N, Sinclair K, Lee S, Gurvich C, Fitzgerald PB, Burger H. Estrogens and men with schizophrenia: is there a case for adjunctive therapy? Schizophr Res. 2011 Feb;125(2-3):278-83. doi: 10.1016/j.schres.2010.10.009. Epub 2010 Nov 9. PMID 21062669
- See also: Centre website — http://www.maprc.org.au/home